CLINICAL TRIAL: NCT06026930
Title: Influence of Low-level Laser Therapy Versus Low-intensity Pulsed Ultrasound on Different Orthodontic Tooth Movements: A Comparative Clinical Investigation
Brief Title: Influence of Low-level Laser Therapy Versus Low-intensity Pulsed Ultrasound on Different Orthodontic Tooth Movements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, farouk ahmed hussein, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 926/91
Record Dates: First submitted 2023-08-19; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Effect of Low Level Laser Versus Low Intensity Pulsed Ultra Sound on Rate of Different Orthodontic Tooth Movement by Millimeter
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Lipus side: canine retraction (Experimental): application of LIPUS with translation of maxillary canine that will be performed on intervention sides according to a standardized protocol
  Interventions: Device: low-level laser therapy
- LIPUS side control side (No Intervention): LIPUS side:canine retraction control side
- LLLT side canine retraction (Experimental): translation of maxillary canine that will be performed with LLLT application according to a standardized protocol
  Interventions: Device: low-level laser therapy
- LLLT side canine retraction control side (No Intervention): LLLT side canine retraction control side wihout intervention
- LIPUS groupMolar distalization group inrervention side (Experimental): distalization assisted with LIPUS according to a standardized protocol
  Interventions: Device: low-level laser therapy
- LIPUS groupMolar distalization group control side (No Intervention): distalization without LIPUS intervention
- LLLT group: distalization intervntion side (Experimental): distalization will be commenced with application of LLLT according to a standardized protocol
  Interventions: Device: low-level laser therapy
- LLLT group: distalization control side (No Intervention): distalization will be commenced without application of LLLT according to a standardized protocol
- LIPUS group: leveling and alignment (Experimental): leveling and alignment assisted with LIPUS according to a standardized protocol
  Interventions: Device: low-level laser therapy
- LLLT group: leveling and alignment (Experimental): leveling and alignment be commenced with application of LLLT according to a standardized protocol
  Interventions: Device: low-level laser therapy
- leveling and alignment without intervention (No Intervention): leveling and alignment without intervention
- LIPUS group: Intrusion (Experimental): intrusion assisted with LIPUS according to a standardized protocol
  Interventions: Device: low-level laser therapy
- LLLT group: Intrusion (Experimental): intrusion assisted with application of LLLT according to a standardized protocol
  Interventions: Device: low-level laser therapy
- intrusion control group (No Intervention): intrusion without intervention

INTERVENTIONS:
Device: low-level laser therapy — LLLT and LIPUS has been found to speed up OTM by stimulating the RANK/RANKL/OPG system to initiate osteoclast formation.
  Other Names: low intensity pulsed ultrasound
  Arms: LIPUS group: Intrusion; LIPUS group: leveling and alignment; LIPUS groupMolar distalization group inrervention side; LLLT group: Intrusion; LLLT group: distalization intervntion side; LLLT group: leveling and alignment; LLLT side canine retraction; Lipus side: canine retraction

SUMMARY:
The aim of this prospective clinical project will be to compare the effect of low-level laser therapy versus low intensity pulsed ultrasound on the rate of different orthodontic tooth movements

DETAILED DESCRIPTION:
The aim of this prospective clinical project will be to compare the effect of low-level laser therapy versus low intensity pulsed ultrasound on the rate of different orthodontic tooth movements, specifically; canine retraction, incisors' leveling and alignment, maxillary molar distalization, and incisors' intrusion

ELIGIBILITY:
Inclusion Criteria:

- A- leveling and alignment Eligibility criteria

1. Age ranges from 14 to 17 years. 2. Bilateral Class II molar relationship. 3. Skeletal Class I or mild Class II relationship. 4. Normal or decreased vertical height. 5. No posterior crowding or spaces. 6. Fully erupted maxillary first and second molars. 7. Congenitally missing or extracted third molars. 8. Good oral hygiene. 9. Absence of any periodontal disease and alveolar bone loss. 10. Absence of medications that may inhibit orthodontic movement

Lower incisor leveling and alignment Inclusion criteria Complete permanent dentition (third molars not included); Moderate mandibular anterior crowding (with little's irregularity index score greater than 4 mm) who required non-extraction approach in the mandibular arch; No tooth size, shape or root abnormalities visible on the patient's radiographic records; No spaces in the mandibular arch; No blocked out tooth that did not allow for placement of the bracket at the

initial bonding appointment; 6. No required management with interproximal stripping, inter-maxillary elastics, open NiTi springs, and removable or extra-oral devices. Canine retraction Eligibility criteria

Age, 15 to 25 years; Class ii division 1 malocclusion with mild or no crowding; No previous orthodontic treatment; No systemic disease that might have affected bone formation or density, such as osteoporosis, hyperparathyroidism, or vitamin d deficiency; Adequate oral hygiene; Probing depth values not exceeding 3 mm across the Entire dentition; Adequate thickness of the attached gingiva (1-2 mm); No radiographic evidence of bone loss

Exclusion Criteria:

- Patients who required surgery to correct skeletal discrepancies. Patients with congenital dentoskeletal disorders. Missed or mutilated teeth in maxillary arch. Patients with poor oral hygiene and/or periodontally compromised patients Severe dental crowding that necessitates an extraction approach 2. Abnormal anteroposterior and vertical relationships; 3. Patients with cleft lip and palate, anomalies, and syndromes; 4. Previous orthodontic 5. Treatment; 6. Regular medications intake that could interfere with otm. -

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Influence of low-level laser therapy versus low-intensity pulsed ultrasound on rate of different orthodontic tooth movements by millimeter | post interventionalal at 6months
  rate of orthodontic tooth movement by millimeter

CONTACTS AND LOCATIONS:
Locations (1):
- AlAzhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Maurya RK, Singh H, Kapoor P, Jain U, Mitra R. Effects of low-level laser and low-intensity pulsed ultrasound therapy on treatment duration and pain perception. J Clin Orthod. 2019 Mar;53(3):154-162. No abstract available. PMID 31009384
- [Result] El-Bialy T, Farouk K, Carlyle TD, Wiltshire W, Drummond R, Dumore T, Knowlton K, Tompson B. Effect of Low Intensity Pulsed Ultrasound (LIPUS) on Tooth Movement and Root Resorption: A Prospective Multi-Center Randomized Controlled Trial. J Clin Med. 2020 Mar 16;9(3):804. doi: 10.3390/jcm9030804. PMID 32188053
- [Result] Qamruddin I, Alam MK, Mahroof V, Karim M, Fida M, Khamis MF, Husein A. Biostimulatory Effects of Low-Intensity Pulsed Ultrasound on Rate of Orthodontic Tooth Movement and Associated Pain, Applied at 3-Week Intervals: A Split-Mouth Study. Pain Res Manag. 2021 May 5;2021:6624723. doi: 10.1155/2021/6624723. eCollection 2021. PMID 34035871